CLINICAL TRIAL: NCT03685422
Title: The Use of Preoperative Virtual Reality to Reduce Anxiety and Pain on Gynaecologic Patients Undergoing Surgery
Brief Title: Preoperative Virtual Reality to Reduce Pain on Gynaecologic Patients Undergoing Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018/2200
Record Dates: First submitted 2018-08-22; First posted 2018-09-26 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Pain, Postoperative; Anxiety
Keywords: Virtual Reality; Pain; Anxiety; Analgesia; Patient satisfaction
MeSH Terms: conditions — Pain, Postoperative; Anxiety Disorders; Pain; Agnosia; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): Patients will be given a VR Gear Headset fitted with a smartphone, and will be offered to choose the calming scenario they wish to experience from a set of predefined scenarios before the surgery. They will be given time to experience VR for up to 25 mins. After the VR session, patients will be given questionnaires, satisfaction with VR, and pain scores.
  After the surgery is completed, patient will be transferred to recovery room. Patients may resume VR session for up to 25 mins. After the use of VR, they will be asked on their satisfaction towards the VR experience, and also fill in questionnaires.
  On the same day of surgery (0-24 hours post-op), patients will be asked to have another two more VR sessions (up to 25 mins per session), with questionnaire filled in after the sessions.
  On the second day and third day of the surgery (48-72 hours post-op), questionnaires will be given.
  All the headsets will be disinfected following the hospital's infection control guideline.
  Interventions: Other: Virtual Reality
- Non Virtual Reality (No Intervention): Before the surgery, only questionnaires and pain scores will be documented. After the surgery is completed, patient will be transferred to recovery room. Only questionnaires and pain scores will be documented.
  On the second day and third day of the surgery (48-72 hours post-op), questionnaires will be given.

INTERVENTIONS:
Other: Virtual Reality — Before surgery, consented patients are given a Virtual Reality headset with pre-installed relaxation apps to choose a preferred scenario. Patient will be asked on their satisfaction on the VR experience after the intervention. Visual analog scale-anxiety (VAS-A), Spielberger State-Trait Anxiety Inventory (STAI) and EQ-5D-3L questionnaires will be conducted during this period.
  Arms: Virtual Reality

SUMMARY:
In the perioperative setting, distraction therapies have been used as a technique to reduce anxiety and pain in the perioperative period. Measures employed in the local restructured hospitals include television, magazines, and newspapers. Tablet-based activity, music and video distraction therapy have also been shown to be useful to reduce preoperative anxiety. The investigators propose a prospective study to implement and evaluate the use of Virtual Reality (VR) in decreasing in anxiety and pain undergoing gynaecological surgery.

In the first phase of study, VR will be administered in 110 female adults undergoing day surgery, same-day-admission or in-patient gynecologic surgery in KKH. The VR will be administered using a Samsung Gear VR3 headset fitted with a smartphone. VR images and sound with calming effect will be delivered to the patients for a short duration of up to 25 minutes. This low-intensity activity offers soothing experience to distract the patients from any pain and anxiety. Second phase of study will randomize 110 female adults undergoing gynecologic surgery. Pain and psychological assessment will be conducted after recruitment, and the group assigned to VR group will navigate the VR environment before and after surgery.

DETAILED DESCRIPTION:
Studies have shown that the majority of patients undergoing selective surgery experience different levels of anxiety. The degree of anxiety is influenced by factors such as patient demographic characteristics, type of surgery, previous experiences with operational procedures, willingness to undergo the proposed intervention, perceived rapport with hospital personnel and personal stress threshold. This anxiety has been shown to be correlated with acute postoperative pain and chronic postsurgical pain, which leads to an increased use of postoperative analgesic, slow recovery, and other maladaptation behaviours in paediatric patient like eating disorders. The link between greater preoperative anxiety and the risk for developing chronic postsurgical pain has been documented in a variety of surgical procedures, including elective abdominal hysterectomy, radical mastectomy, breast cancer surgery, and arthroscopic knee surgery. While pharmacological interventions such as opioid-based analgesic are available, other methods to manage anxiety and distract patients from stressors - such as music, television, and virtual reality - have become more popular in the recent years due to their safety, low cost and effectiveness in improving overall patient experience and outcome.

Virtual reality (VR) is a promising new technology that offers opportunities to modulate pain experience and cognition. Patients received VR treatment reported a reduction in pain and anxiety, faster wound healing, decreased chronic pain intensity and other neurorehabilitation improvements. The recent advent of inexpensive consumer VR system has also made VR more accessible to the mass, especially those by Samsung available locally. In SingHealth, VR has been used in neurosurgery for individualized surgery planning for patients with brain tumours, vascular malfunction and skull based tumours. However, there has been little done to investigate the effectiveness of VR during the preoperative period especially in local setting. Therefore, the investigators will investigate the feasibility and practicability of employing VR in anxiety and pain management in patients undergoing same day admission or day surgery. The proposed intervention may not only be implemented in the preoperative environment but also be in other settings such as before diagnostic screening or minor treatments done during inpatient stay or outpatient visit. The use of VR is suitable for those who are preparing for procedures in clinic or ward as an alternative anxiety management without prolonging the preparation time.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants who are ASA 1 & 2 (with well-controlled medical problems)
* Undergo day surgery or same-day -admission gynecologic surgery
* Have no visual impairment

Exclusion Criteria:

* Patients with significant respiratory disease and obstructive sleep apnea
* Patient who are unable to understand questionnaire
* Obstetric patients
* Patients with motion sickness in 3D environment

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only females undergoing gynecologic surgery in KKH will be recruited
Enrollment: 220 (Estimated)
Dates: Start 2019-03-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Pain scores as assessed by Numeric Rating Scale in both groups | 3 days (post-op Day 1-3)
  Difference in pain scores between virtual reality (VR) and non-VR groups. Pain scores (on a numeric rating scale 0-10) will be given to patients, with 0 being no pain and 10 being the worst pain possible.
Quality of recovery as assessed by Quality of Recovery -40 (QoR-40) score in both groups | 3 days (post-op Day 1-3)
  Difference in QoR-40 between virtual reality (VR) and non-VR groups. The QoR-40 is a global measure of quality of recovery. It incorporates five dimensions of health: patient support, comfort, emotions, physical independence, and pain; each item is graded on a five-point Likert scale. QoR-40 scores range from 40 (extremely poor quality of recovery) to 200 (excellent quality of recovery).

SECONDARY OUTCOMES:
Total consumption of morphine in both groups | 3 days (post-op Day 1-3)
  Difference in Morphine (in milligrams) used after surgery between virtual reality (VR) and non-VR groups.
Change in Patient satisfaction as assessed by ordinal scale (VR group only) | 4 days (before surgery till post-op Day 1-3)
  Patients assigned to VR group will be asked on their satisfaction level before and after the use of VR based on ordinal scale (excellent, good, fair, poor).
Visual analog scale-anxiety (VAS-A) score in both groups | 4 days (before surgery till post-op Day 1-3)
  VAS-A score will be collected before and after surgery to assess patients' level of anxiety in both VR and non-VR groups. VAS-A scores from 0 to 10, with 0 being no anxiety and 10 being the greatest anxiety. Higher score indicates a greater level of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Ban Leong Sng, MBBS, MMED, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan JJI, Yeam CT, Kee HM, Tan CW, Sultana R, Sia ATH, Sng BL. The use of pre-operative virtual reality to reduce anxiety in women undergoing gynecological surgeries: a prospective cohort study. BMC Anesthesiol. 2020 Oct 9;20(1):261. doi: 10.1186/s12871-020-01177-6. PMID 33036555

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/22/NCT03685422/Prot_SAP_000.pdf